CLINICAL TRIAL: NCT06745453
Title: Erector Spinae Plane Block for Acute Back Pain in the Emergency Department
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Rush University Medical Center (Other)
Responsible Party: Principal Investigator, Michael Gottlieb, Professor of Emergency Medicine, Rush University Medical Center
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 24062802
Record Dates: First submitted 2024-12-17; First posted 2024-12-20 (Actual); Last update posted 2025-03-10 (Actual); Status verified 2025-03

CONDITIONS: Low Back Pain
Keywords: erector spinae plane block; emergency department; low back pain; regional anesthesia; nerve block
MeSH Terms: conditions — Low Back Pain; Emergencies

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Erector Spinae Plane Block (Experimental): This group will receive the erector spinae plane block
  Interventions: Procedure: Erector Spinae Plane Block
- Sham Procedure (Sham Comparator): This group will receive a sham injection.
  Interventions: Procedure: Sham Procedure

INTERVENTIONS:
Procedure: Erector Spinae Plane Block — Erector Spinae Plane Block
  Arms: Erector Spinae Plane Block
Procedure: Sham Procedure — Sham Procedure
  Arms: Sham Procedure

SUMMARY:
The goal of this clinical trial is to learn if an erector spinae plane block (ESPB; a type of nerve block) works to reduce pain in adults presenting to the emergency department with low back pain. It will also learn if the ESPB reduces pain, disability, and return to work at 7 days. The main questions it aims to answer are:

1. Does the ESPB reduce short-term pain in participants with low back pain?
2. Does the ESPB reduce longer-term pain, reduce disability, and improve return to work and activities in participants with low back pain?

Researchers will compare ESPB to a placebo (an injection that does not involve a nerve block) to see if ESPB works to treat low back pain.

Participants will:

Receive either the ESPB or a placebo injection in the emergency department Report their pain scores for up to 120 minutes Report their pain, disability, and return to work at 7 days

ELIGIBILITY:
Inclusion Criteria:

* Adults (age ≥18 years) presenting to the emergency department with isolated low back pain present less than 6 total weeks.

Exclusion Criteria:

* Do not speak English or Spanish as a primary language
* Are incarcerated
* Have a known pregnancy
* Are allergic to amide-type local anesthetics
* Are unable to tolerate positioning for the procedure
* Have a critical illness precluding the ability to perform the procedure.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 62 (Estimated)
Dates: Start 2025-02-03 (Actual); Primary Completion 2026-06-23 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Pain score at 120 minutes post-intervention as assessed using a 10-point numeric rating scale | Change from baseline to 120 minutes post-intervention
  Zero is equivalent to no pain and 10 indicates worst pain imaginable

SECONDARY OUTCOMES:
Pain score at 30 minutes post-intervention as assessed using a 10-point numeric rating scale | Change from baseline to 30 minutes post-intervention
  Zero is equivalent to no pain and 10 indicates worst pain imaginable
Pain score at 60 minutes post-intervention as assessed using a 10-point numeric rating scale | Change from baseline to 60 minutes post-intervention
  Zero is equivalent to no pain and 10 indicates worst pain imaginable
Degree of disability assessed via the Roland-Morris disability questionnaire at 7 days | Assessed as the change in Roland-Morris disability questionnaire scores between baseline and 7 day follow up
  Participants will be scored using the validated Roland-Morris disability questionnaire.
Pain score at 7 days post-intervention as assessed using a 10-point numeric rating scale | Pain score assessed at 7 days post-intervention
  Zero is equivalent to no pain and 10 indicates worst pain imaginable
Opioid medications taken in the 7 days following the intervention | Measured at 7 days post-intervention
  Calculated in morphine milligram equivalents
Follow up visits related to low back pain in the 7 days following the intervention | Assessed at 7 days
  Based upon patient self-report
Return to work and activities assessed via the Work Productivity and Activity Impairment Questionnaire: General Health version 2.0 | Assessed at 7 days
  Assessed using the validated Work Productivity and Activity Impairment Questionnaire: General Health version 2.0 questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Michael Gottlieb, MD, Principal Investigator — Rush University Medical Center
Locations (1):
- Rush University Medical Center, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: No